CLINICAL TRIAL: NCT06116851
Title: Prostate Metabolism, Cancer Risk and Gut Microbiota
Acronym: PROMIC
Status: Recruiting | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Collaborators: University of Turku (Other)
Responsible Party: Sponsor
Other Study IDs: 15/1801/2022
Record Dates: First submitted 2023-04-14; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Prostate Cancer; Prostate Hyperplasia
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Hyperplasia | interventions — Magnetic Resonance Spectroscopy; Blood Specimen Collection; Urination; Transurethral Resection of Prostate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Blood and urine samples: Serum, plasma and whole blood samples will be collected to measure steroid hormone concentrations, global analysis of molecular lipids and polar metabolites, and for DNA sequence analysis.
  2. Stool samples:Stool samples will be collected and stored in OMNImetGUT and OMNIgeneGUT and eSwab tubes. Samples will be used for sequencing and for antimicrobial susceptibility testing.
  3. Tissue samples: Fresh frozen tissue samples will be collected from subjects going to surgery (TURP, RALP, Cystoprostatectomy) for sequencing and mass spec analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- suspicion: Inclusion criteria for the suspicion cohort include clinical suspicion for PCa and indication for PCA diagnostics based on any of the following: 1) elevated PSA (>2.5 ng/ml), 2) palpable prostate tumor/nodule, 3) image finding suggestive of PCa.
  The suspicion cohort will include a total of 300 subjects who will undergo PCa diagnostics including prostate MRI, and transrectal ultrasound (TRUS) guided prostate biopsies. After the diagnostic procedures all subjects are categorized to one of the following groups: 1) subject without PCa, 2) subject with clinically non-significant PCa (ISUP grade 1/Gleason 3+3), 3) clinically significant PCa (ISUP grade >1/>Gleason 3+3).
  Based on the outcome of the PCa diagnostics and planned clinical treatment, subjects may be eligible to other cohorts as well.
  Interventions: Other: MRI scan and laboratory visit; Procedure: Prostate biopsies
- cancer (radical prostatectomy) cohort: Inclusion criteria for the cancer cohort include clinically significant prostate cancer planned to be treated with radical prostatectomy with or without pelvic lymph node dissection. The cancer cohort will include a total of 50 subjects.
  Interventions: Procedure: Radical prostatectomy and blood, urine and tissue sampling
- benign/TURP-cohort: Inclusion criteria for the benign (TURP) cohort includes benign prostate hyperplasia (BPH) planned to be treated with transurethral resection of the prostate (TURP). The benign/TURP-cohort will include a total of 50 subjects.
  Interventions: Procedure: TURP and blood, urine and tissue sampling
- benign/cystectomy: Inclusion criteria for the benign/cystectomy cohort includes bladder cancer planned to be treated with removal of the urinary bladder and prostate (cystoprostatectomy). The benign/cystectomy cohort will include a total of 25 subjects.
  Interventions: Procedure: Radical cystoprostatectomy and blood, urine and tissue sampling

INTERVENTIONS:
Other: MRI scan and laboratory visit — Prostate MRI scan is performed according to the protocol used in earlier studies (PMID 31158230). In addition to the PCa diagnostics, the scan will include abdominal imaging to body composition analysis (visceral and subcutaneous fat and psoas muscle). Baseline blood and urine samples are collected in Turku University Hospital laboratory.
  Groups: suspicion
Procedure: Prostate biopsies — The visit follows routine outpatient clinic protocol. The results from MRI and laboratory findings are discussed and the potential benefits and harms from prostate biopsies are evaluated. After a mutual decision, prostate biopsies are performed.
  Groups: suspicion
Procedure: Radical prostatectomy and blood, urine and tissue sampling — Baseline blood and urine samples are collected at the time of surgery. Robotic assisted laparoscopic prostatectomy (RALP) is performed according to routine protocol. Routine diagnostic histopathological procedures will be followed, and study tissue samples are obtained in the department of pathology.
  Groups: cancer (radical prostatectomy) cohort
Procedure: TURP and blood, urine and tissue sampling — Baseline blood and urine samples are collected the time of surgery. TURP is performed according to normal protocol. Routine diagnostic histopathological procedures will be followed in the department of pathology. Additionally, tissue samples (a total of 10 resection chips) will be collected for study analyses. Due to the study, no additional tissue samples are removed, i.e. study samples are from the tissues removed as clinically indicated.
  Groups: benign/TURP-cohort
Procedure: Radical cystoprostatectomy and blood, urine and tissue sampling — Baseline blood and urine samples are collected at the time of surgery. Radical cystoprostatectomy is performed according to routine protocol. Routine diagnostic histopathological procedures will be followed, and study tissue samples are obtained in the department of pathology.
  Groups: benign/cystectomy

SUMMARY:
This is a prospective, single center translational multiple cohort study to investigate the association of gut microbiota and prostate cancer.

DETAILED DESCRIPTION:
Prostate cancer (PCa) is a significant health care system challenge. PCa is the most common male cancer in Finland and most western countries. Interestingly, although the incidence of indolent (latent) PCa is very similar throughout the globe, there is a remarkable global age-adjusted incidence variation (up to 40-fold difference between highest and lowest incidences).

Epidemiological data suggest that aging in men is associated with neoplastic processes in the prostate but only a subset of men will develop a true malignancy potentially affecting their life-span or quality of life. Genetic factors have a significant effect on PCa risk, but very likely life-style (e.g. diet and physical activity) affect PCa risk as well, but the mechanisms mediating protective or harmful effects of life-style remain unclear.

Gut microbiota, i.e. the collection of microbes colonizing the gastrointestinal tract, has been acknowledged to play significant role in many metabolic pathways and pathogenetic processes in the human body. Although there is some evidence suggesting that gut microbiota affects therapy responses (especially androgen deprivation) in PCa, it´s potential role in prostate carcinogenesis is not well documented. Our previous studies suggest that gut microbiota composition is different in men with and without PCa potentially contributing to the Pca risk, and that changes in steroid hormone synthesis may be one mechanism how gut microbiota affects PCa risk.

PROMIC is a prospective, single center translational multiple cohort study to investigate the association of gut microbiota and PCa. The main aim is to validate our preliminary findings of association between gut microbiota and PCa. We also study metabolic characteristics in the gut, systemic circulation, and prostate tissue in men with different gut microbiota signatures. The study is carried out in Turku University Hospital and University of Turku.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form.
* Ability and stated willingness to comply with all study procedures and availability for the duration of the study.

Exclusion Criteria:

* inability to comply with study procedures or unwillingness to participate in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Suspicion cohort: cohort include clinical suspicion for PCa and indication for PCA diagnostics based on any of the following: 1) elevated PSA (>2.5 ng/ml), 2) palpable prostate tumor/nodule, 3) image finding suggestive of PCa.
  Cancer cohort, (RALP): cohort include clinically significant prostate cancer planned to be treated with radical prostatectomy with or without pelvic lymph node dissection.
  TURP cohort: cohort includes benign prostate hyperplasia (BPH) planned to be treated with transurethral resection of the prostate (TURP).
  Cystectomy cohort: cohort includes bladder cancer planned to be treated with removal of the urinary bladder and prostate (cystoprostatectomy).
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-01-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Gut microbiota signature | immediately before prostate biopsy
  Gut microbiota signature in men with clinically significant prostate cancer, clinically non-significant prostate cancer, and benign prostate histology

SECONDARY OUTCOMES:
Gut metabolomics | immediately before prostate biopsy
  Metabolic characteristics in the gut in men with different gut microbiota signatures

OTHER OUTCOMES:
Systemic circulation metabolomics | immediately before prostate biopsy
  Metabolic characteristics in the systemic circulation in men with different gut microbiota signatures
Prostate tissue metabolomics | immediately before prostate biopsy
  Metabolic characteristics in the prostate tissue in men with different gut microbiota signatures

CONTACTS AND LOCATIONS:
Overall Officials: Peter J. Bostrom, MD, PhD, Principal Investigator — Turku University Hospital and University of Turku
Locations (2):
- Finland (2):
  - University of Turku, Turku
  - Turku University Hospital, Turku